CLINICAL TRIAL: NCT07218198
Title: A Stepped Wedged, Cluster Randomized Clinical Trial to Evaluate the Efficacy of a Clinical Decision Support Tool in the Treatment of Uncontrolled Hypertension
Brief Title: Clinical Decision Support Tool for the Treatment of Uncontrolled Hypertension
Acronym: AI-HTN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V2.0 11Dec2025
Record Dates: First submitted 2025-10-14; First posted 2025-10-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Hypertension (HTN); Blood Pressure, High; Blood Pressure Control
Keywords: Uncontrolled Hypertension; Hypertension; Blood Pressure; High Blood Pressure; Artificial Intelligence; AI
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The study is a stepped wedge cluster randomized trial. All participating clinicians will receive access to the CDS tool, but clinicians will have different start dates for the tool.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care for Hypertension Management (Active Comparator): Clinicians will use their own standard of care recommendations for combinations of medications.
  Interventions: Other: Standard medical treatment
- Clinical Decision Support Tool (Experimental): Clinical Decision Support Tool embedded into the Electronic Medical Record to help support clinicians to prescribe more effective combinations of medications
  Interventions: Other: Clinical Decision Support Tool

INTERVENTIONS:
Other: Standard medical treatment — Clinicians will use their own standard of care recommendations for combinations of medications.
  Other Names: hypertension; hypertension management
  Arms: Standard of Care for Hypertension Management
Other: Clinical Decision Support Tool — Clinical Decision Support Tool embedded into the Electronic Medical Record to help support clinicians to prescribe more effective combinations of medications
  Other Names: hypertension; hypertension management
  Arms: Clinical Decision Support Tool

SUMMARY:
The goal of this clinical trial is to study whether having a clinical decision support (CDS) tool available to clinician use will more effectively lower BP 4 weeks after an outpatient visit compared with usual care. The main objective is to assess the impact of the CDS tool, that is embedded with the electronic medical record (EMR), that is available during outpatient clinical encounters, on blood pressure (BP) changes among participants with uncontrolled hypertension.

Participants will:

Visit the clinic 4 weeks, after their initial clinician visit, for a BP check.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years of age or older
2. Electronic Health Record (EHR) of hypertension AND prescribed at least one BP lowering medication
3. Office systolic BP of 130 mmHg or higher
4. Willing and able to comply with the study instructions AND attend a scheduled study visit

Exclusion Criteria:

1. Women who are pregnant, plan to become pregnant, or are breast-feeding
2. Know heart failure with reduced ejection fraction and a left ventricular ejection fraction of less than 40%
3. End-stage kidney disease currently undergoing renal replacement therapy, or an eGFR < 15ml/min/1.73m2
4. In the opinion of the investigator, any other condition that will preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic automated office blood pressure (AOBP) | 4 weeks
  Clinical Decision Support (CDS) Tool is available, Change from baseline in systolic automated office blood pressure (AOBP) at 4 weeks.

SECONDARY OUTCOMES:
Change in diastolic automated office blood pressure (AOBP) | 4 weeks
  Percentage of Participants with controlled BP (<130mmHg), Change from baseline in diastolic automated office blood pressure (AOBP) at 4 weeks.

OTHER OUTCOMES:
Safety of the CDS Tool | 4 weeks
  Number of participants with treatment related adverse events, Change from baseline at 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Laffin, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Result] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):1269-1324. doi: 10.1161/HYP.0000000000000066. Epub 2017 Nov 13. No abstract available. PMID 29133354
- [Result] Mroz T, Griffin M, Cartabuke R, Laffin L, Russo-Alvarez G, Thomas G, Smedira N, Meese T, Shost M, Habboub G. Predicting hypertension control using machine learning. PLoS One. 2024 Mar 20;19(3):e0299932. doi: 10.1371/journal.pone.0299932. eCollection 2024. PMID 38507433
- [Result] Darricarrere C, Jacquot E, Bricout S, Louis C, Benard M, Poulter NR. Uncontrolled blood pressure and therapeutic inertia in treated hypertensive patients: A retrospective cohort study using a UK general practice database. J Clin Hypertens (Greenwich). 2023 Oct;25(10):895-904. doi: 10.1111/jch.14699. Epub 2023 Sep 22. PMID 37740433